CLINICAL TRIAL: NCT05427981
Title: Functional Brain Mechanisms Underlying the Anti-Suicidal Effects of Low-dose Buprenorphine in Major Depression
Brief Title: Anti-suicidal Effects of Buprenorphine In Depressed Individuals
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: U.S. Department of Health and Human Services OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. This study will not resume recruitment after the resumption of research.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Mina.Rizk, Assistant professor, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #8086
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Suicidal Ideation; Major Depressive Disorder
MeSH Terms: conditions — Suicidal Ideation; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Buprenorphine (Experimental): Buccal Films
  Interventions: Drug: Belbuca Buccal Product
- Placebo (Placebo Comparator): Buccal Films
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Belbuca Buccal Product — Buprenorphine Buccal Films
  Arms: Buprenorphine
Other: Placebo — Placebo Buccal Films
  Arms: Placebo

SUMMARY:
This study aims to examine the effect of low-dose buprenorphine as an add-on to treatment-as-usual for suicidal ideation in individuals with major depression, and investigate the functional brain activity related to its potential anti-suicidal effect.

DETAILED DESCRIPTION:
Buprenorphine is an approved treatment for pain and opioid relapse prevention. Buprenorphine has recently shown promise in the treatment of depression and suicidal ideation relatively faster than currently available antidepressants, but its mechanisms in treating these conditions are unknown. Buprenorphine activates the mu opioid receptor in the brain and blocks the kappa opioid receptor. Activation of the mu receptors produces pleasant emotions while the kappa receptors are linked to dysphoria and other negative emotional states. By blocking kappa receptors, buprenorphine may reduce negative emotions and improve suicidal thoughts.

In this project, we will compare buprenorphine to placebo as adjunctive to usual treatments for patients who still have depression and suicidal thoughts despite being treated with adequate antidepressant medications for at least 4 weeks. We hypothesize that suicidal ideation will decrease after two weeks of treatment in the buprenorphine group relative to the placebo group.

Using functional magnetic resonance imaging, we will also examine the effects of buprenorphine on the activity of brain regions involved in the brain's response to negative emotions and test whether these effects are associated with the reduction in suicidal thoughts. This would provide some evidence that the antidepressant and anti-suicidal effects of buprenorphine are related to its kappa opioid receptor blockade.

The mechanism of action of buprenorphine is different from the currently available antidepressants. This study will help understand this mechanism which may help refine the use of buprenorphine in this context. Research in this area may also facilitate the development of new anti-suicidal treatments (i.e., other opioid-active compounds).

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female.
4. Aged 18-65 years.
5. Ability to take oral medication and be willing to adhere to the treatment regimen.
6. Current major depressive episode.
7. Hamilton Depression Rating Scale (HDRS) Score > 16.
8. Active suicidal ideation (Columbia Suicide Severity Rating Scale (C-SSRS) of 3 or more).
9. Participants must have been on a medication regimen for depression that includes an adequate dose of antidepressant for at least the past 4 weeks.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Current active psychosis or mania.
2. Current or past alcohol use disorder or substance use disorder involving any prescribed or any illicit drug (opioid, benzodiazepine, or other drug use) including mild severity.
3. Family history of alcohol or substance use disorder in a first-degree relative.
4. Current or past history of prescription or non-prescription opioid use.
5. History of other risk factors for the development of opioid misuse and opioid use disorder other than comorbid depression (e.g., homelessness, criminal record, aggressive or violent behavior that resulted in injury to another person).
6. Current acute or chronic pain.
7. Neurological disorders (e.g., epilepsy, brain tumors or patients with increased intracranial pressure due to other reasons).
8. A history of prior head trauma with evidence of cognitive impairment. Participants who endorse a history of prior head trauma will be administered the Trail-making A and B test. Those who score 1.5 standard deviations below the mean on the Trail-making A or B will be excluded from study participation.
9. Active significant medical illness that would make study participation hazardous to the participant or compromise study findings or would prevent the participant from completing the study (e.g., oral mucositis, orthostatic hypotension, history of hypotensive disorders, hypokalemia, hypomagnesemia, or clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, or active myocardial ischemia, history of Long QT syndrome or immediate family member with this condition, moderate to severe hepatic impairment or hepatitis, liver cirrhosis , severe chronic pulmonary diseases, significant respiratory depression, acute or severe bronchial asthma, known or suspected gastrointestinal obstruction, including paralytic ileus).
10. Participants taking medications that prolong the QT interval (e.g., Class IA antiarrhythmic medications (e.g., quinidine, procainamide, disopyramide) or Class III antiarrhythmic medications (e.g., sotalol, amiodarone, dofetilide)).
11. Participants taking medications with potentially clinically-significant drug interactions with BELBUCA , including benzodiazepines, central nervous system (CNS) depressants (e.g., alcohol, anxiolytics, general anaesthetics, hypnotics, neuroleptics, phenothiazines, sedatives, tranquilizers), other opioid analgesics, muscle relaxants, diuretics, anticholinergic drugs, non-nucleoside reverse transcriptase inhibitors (e.g., efavirenz, nevirapine, etravirine, delavirdine), protease inhibitors (e.g., atazanavir, ritonavir). Additionally, patients must discontinue CYP3A4 strong inhibitors (e.g., clarithromycin, telithromycin, nefazodone, itraconazole, ketoconazole) 2 weeks before initiation of the study.
12. Known allergy or sensitivity to buprenorphine.
13. If female, pregnancy, abortion or miscarriage in the previous two months, current breastfeeding or plans to conceive during the course of study participation. Patients who are not on contraceptives will be asked to at least use barrier methods during sexual intercourse. All patients must commit to not attempting to become pregnant during participation in the study.
14. Inability to read and speak English fluently.
15. Metal implants or paramagnetic objects contained within the body (including heart pacemaker, shrapnel, or surgical prostheses) which may present a risk to the subject or interfere with the MR scan, according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects", F. G. Shellock, Lippincott Williams and Wilkins NY 2001. Additionally, transdermal patches will be removed during the MRI.
16. Claustrophobia significant enough to interfere with MRI scanning.
17. Weight over 350 lbs or inability to fit into MRI scanner.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-01-14 (Estimated); Study Completion 2024-01-14 (Estimated)

PRIMARY OUTCOMES:
Changes in Beck Scale for Suicidal Ideation (SSI) scores from pre- to Week 2 post-treatment. | 2 Weeks
  Clinician-based questionnaire measuring level of suicidal ideas over the last 7 days; 21 items scored 0 to 2; total score ranges from 0 to 38 (last 2 items not counted), higher scores mean more intense suicidal ideas.

SECONDARY OUTCOMES:
Changes in functional magnetic resonance imaging (fMRI) blood oxygen- level dependent (BOLD) signal in the amygdala in response to negative vs. neutral pictures from pre- to Week 2 post-treatment | 2 Weeks
  fMRI negative picture task administered at baseline and week 2 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mina M Rizk, MD, Principal Investigator — New York State Psychiatric Institute; Jeffrey M Miller, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No